CLINICAL TRIAL: NCT06963827
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate Efficacy and Safety of Mezagitamab (TAK-079) in Study Participants With Primary IgA Nephropathy in Combination With Stable Background Therapy
Brief Title: A Study of Mezagitamab in Adults With Primary IgA Nephropathy Kidney Condition
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-079-3001; 2025-520825-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Kidney Disease
Keywords: TAK-079; Drug Therapy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mezagitamab (Experimental): Participants will receive mezagitamab injections, subcutaneously (SC), for approximately 22 weeks in each 52-week period.
  Interventions: Drug: Mezagitamab
- Placebo (Placebo Comparator): Participants will receive mezagitamab-matching placebo injections, SC for approximately 22 weeks in each 52-week period.
  Interventions: Drug: Placebo
- Open-label Mezagitamab (Experimental): Participants will receive mezagitamab injections, SC for approximately 22 weeks in each 52-week period.
  Interventions: Drug: Mezagitamab

INTERVENTIONS:
Drug: Mezagitamab — Mezagitamab injections administered SC.
  Other Names: TAK-079
  Arms: Mezagitamab; Open-label Mezagitamab
Drug: Placebo — Mezagitamab-matching placebo injections administered SC.
  Arms: Placebo

SUMMARY:
Immunoglobulin A nephropathy (IgAN) is a kidney condition. It happens when the body's immune system creates groups of proteins (called immune complexes) that build-up in the kidneys causing swelling (inflammation). Over time, this inflammation may lead to kidney damage and cause the kidneys to no longer work properly. The main aim of this study is to check how well mezagitamab changes protein levels in the urine (proteinuria) compared to placebo in adults with primary IgAN. A placebo looks like medicine but doesn't have any active ingredients in it. Other aims are to check how safe mezagitamab is and how well participants with primary IgAN can tolerate it compared to placebo, and to find out if and how well mezagitamab continues to maintain kidney function over the long term compared to placebo.

Participants will be placed in 1 of the 2 treatment groups; the main group and the open-label group. In the main group, participants will be placed in 1 of the 2 treatment groups by chance (either mezagitamab or placebo) at a 2:1 ratio. This means that out of 3 participants, 2 will receive mezagitamab and 1 will receive placebo. The participants will receive either mezagitamab or placebo for almost half a year in two 1-year cycles. They will be observed for another half year in each 1-year cycle and will have check-ups about every month during this time.

In the open-label group, a small number of participants who have lower levels of protein in their urine or have kidneys that do not filter the blood well, will receive mezagitamab treatment. This will include participants who have previously received mezagitamab in another study, TAK-079-1006. Every participant will receive mezagitamab in the same way as those in the main group receiving mezagitamab.

During the study, participants will visit their study clinic several times.

ELIGIBILITY:
* Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Either UPCR greater than or equal to (≥) 0.8 gram per gram (g/g) or urine protein excretion (UPE) ≥1 grams per day (g/day), calculated from a 24-hour urine collection during the screening period (only applicable for the main group).
2. eGFR greater than (>)30 milliliters per minute per 1.73 meter square (mL/min/1.73m^2) at screening based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (only applicable for the main group).
3. No prior exposure to anti- cluster of differentiation 38 (CD38) therapy period (only applicable for the main group).
4. The participant is at least aged 18 years or the local legal age if greater than 18 years, inclusive.
5. The participant (and the participant's legally acceptable representative, if applicable per local regulations or determination) has provided informed consent (that is, in writing, documented via a signed and dated informed consent form [ICF]) and any required privacy authorization before the initiation of any clinical trial procedures.
6. Renal biopsy report supporting diagnosis of primary IgAN within 10 years before signing informed consent for the clinical trial. The redacted report must be made available for review. A renal biopsy may be performed during screening.
7. Participants must be on stable renin-angiotensin-aldosterone system (RAAS) inhibitor therapy with an angiotensin-converting enzyme inhibitor (ACE-I) and/or angiotensin receptor blocker (ARB) or endothelin receptor antagonist (ERA) or mineralocorticoid receptor antagonist (MRA) agent for at least 12 weeks before signing the ICF with dosing at the maximally tolerated or labeled dose as determined by the investigator, with the intent to continue stable dosing during the clinical trial. Those intolerant of RAAS inhibitor therapy are potentially eligible after consultation with the medical monitor. Intolerance is defined as a documented side effect causing discontinuation of the therapy.
8. Women of childbearing potential who are not pregnant during screening (confirmed by negative serum human chorionic gonadotropin [hCG]) and on Visit 1 before first dose of trial intervention (confirmed by negative urine pregnancy test).
9. Any one of the following (only applicable for the open-label cohort):

   1. Participants in Study TAK-079-1006 who completed the Week 96 visit or the retreatment period with either UPCR >0.5 g/g or UPE >0.5 g/d calculated from a 24-hour urine collection during the screening period and eGFR >30 mL/min/1.73m^2 at screening based on the CKD-EPI formula.
   2. UPCR <0.8 g/g and UPE ≥0.75 and <1.0 g/day, by 24-hour urine collection during the screening period and eGFR > 30 mL/min/1.73m^2 at screening based on the CKD-EPI formula.
   3. UPCR ≥ 0.8 g/g or UPE ≥ 1.0 g/d by 24-hour urine collection during the screening period and eGFR ≥25 and ≤30 mL/min/1.73m^2 at screening based on the CKD-EPI formula.

      * Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. Kidney biopsy exhibiting significant concomitant renal disease other than IgAN (for example, diabetic nephropathy, lupus nephritis, minimal change disease).
2. Secondary IgAN (such as with significant liver disease, immunoglobulin A (IgA) vasculitis, inflammatory bowel disease, and seronegative spondyloarthropathies).
3. Evidence of rapidly progressive glomerulonephritis (loss of ≥50% of eGFR within 3 months before the signing of the ICF).
4. Diagnosis of nephrotic syndrome defined as 24-hour proteinuria >3.5 g/day or hypoalbuminemia (<3.0 grams per deciliter [g/dL]) with or without peripheral edema.
5. Renal or other organ transplantation prior to or expected during the clinical trial.
6. Treatment with oral immunosuppressive agents (including cyclophosphamide, mycophenolate mofetil, cyclosporine, azathioprine, calcineurin inhibitors) or biologic therapy for immunomodulation (including immunomodulatory monoclonal or polyclonal antibodies) within 6 months (both B-cell and non-B-cell directed agents) before signing of the ICF.
7. If the participant has received anti-CD20 treatment, the participant is excluded if either of the following apply:

   1. The last dose was received within 6 months before the signing of the ICF.
   2. The last dose was received between 6 and 12 months before the signing of the ICF and the participant has a CD19+ count below the lower limit of normal.

   Note: Participants who have received the last dose of anti-CD20 treatment >12 months before the signing of the ICF are not excluded from clinical trial participation based on this criterion and are not required to undergo CD19+ testing.
8. Use of systemic corticosteroids at an average dose of 40 milligrams (mg) prednisone equivalent or higher for more than 14 days within 4 months of the screening visit, or use of oral budesonide delayed release capsules within 1 year of the screening visit.
9. The participant has received a live or live-attenuated vaccine within 4 weeks before signing the ICF or has any live or live-attenuated vaccine planned during the clinical trial.
10. Participation in any other investigational drug trial (including vaccine trial) with receipt of at least 1 dose of investigational drug, or has been exposed to another investigational agent within 4 weeks or 5 half-lives, whichever is longer, before Visit 1.
11. The participant has active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
12. The participant has had any of the following types of infections within the specified timeframes where applicable:

    1. Active bacterial, viral, fungal infection (except for the common cold and onychomycosis), or any other serious infection within 2 weeks of signing the ICF. Any anti-infective course for infection must be completed at least 2 weeks before Visit 1.
    2. Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) infection within 4 weeks of signing the ICF.
    3. Opportunistic infection or treatment for an opportunistic infection lesser than or equal to (≤)12 weeks before signing the ICF.
13. In the opinion of the investigator, the participant is currently experiencing any medical condition that might interfere with participation in the trial (for example, significant ocular, cardiovascular, pulmonary, hematologic, gastrointestinal, endocrinologic, hepatic, renal, neurologic, malignancy, infectious disease, immunodeficiency, or alcohol and drug abuse), that poses an added risk for the participant or could confound the assessment of trial results.
14. In the opinion of the investigator, the participant has a serious medical or psychiatric illness that could potentially interfere with the completion of treatment.
15. The participant has a history of major surgery within 3 months before screening (or longer, at the discretion of the investigator); or, either has a planned tonsillectomy or underwent a tonsillectomy within 6 months before screening.

    Note: Major surgery typically requires at least 1 night in the hospital.
16. History of malignancy (including myelodysplastic syndrome) within 5 years of signing the ICF, except for adequately treated non-melanoma skin cancer, superficial bladder cancer, and curatively treated cervical carcinoma-in-situ.
17. The participant has a history of a severe allergic or anaphylactic reaction to recombinant proteins or excipients used in the mezagitamab or placebo formulation.
18. The participant has (1) been diagnosed with or has suspected chronic obstructive pulmonary disease (COPD) or asthma and (2) has a prebronchodilatory forced expiratory volume in 1 second (FEV1) <50% of predicted normal at screening.
19. The participant is capable of breastfeeding but does not agree to forego breastfeeding from first dose of investigational medicinal product (IMP) through 30 days after the last dose of IMP.
20. The participant is an individual with potential for pregnancy but does not agree to use at least 1 form of highly effective contraception and 1 barrier method of contraception (preferably male condom) when engaging in heterosexual sex for the protocol specified duration after the last dose of IMP.
21. The participant is a sexually active, non-sterilized individual who produces sperm but does not agree to use a barrier method (preferably male condom) combined with at least 1 form of highly effective contraception for any partner(s) with potential for pregnancy when engaging in heterosexual sex for the protocol specified duration after the last dose of IMP.
22. In the investigator's opinion, the participant (and the participant's legally acceptable representative, if applicable per local regulations or determination) is unwilling and/or unable to understand and fully comply with clinical trial procedures and requirements (including digital tools and applications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-09-07 (Estimated); Study Completion 2030-01-14 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Proteinuria at Week 36 | From Baseline to Week 36
  Proteinuria will be assessed by urine protein to creatinine ratio (UPCR) calculated from a 24-hour urine collection.

SECONDARY OUTCOMES:
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52 and 104, Respectively | From Baseline to Weeks 52 and 104
The Rate of Change in eGFR From Baseline at Weeks 52 and 104, Respectively | From Baseline to Weeks 52 and 104
  The rate of change in eGFR from baseline is measured as eGFR total slope.
Time from Baseline to the First Occurrence of Any of the Pre-specified Kidney Failure Composite Assessment Criteria | From Baseline to Week 104
  The pre-specified assessment criteria will include: sustained decline in eGFR of ≥30% from baseline over at least 4 weeks; sustained eGFR <15 mL/min/1.73 m^2 over at least 4 weeks; initiation of maintenance dialysis defined as dialysis performed for at least 4 weeks; receipt of kidney transplant; or death from kidney failure. Time from baseline to first occurrence of any of the above assessment criteria would be reported.
Change from Baseline in Proteinuria Levels at Week 104 | From Baseline to Week 104
  Proteinuria will be assessed by UPCR calculated from a 24-hour urine collection.
Resolution of Hematuria at Weeks 36, 52 and 104, Respectively | Weeks 36, 52 and 104
  Resolution of hematuria is defined as having a negative hematuria result at the specified visit among those participants with positive hematuria at Baseline.
Number of Participants With Antidrug Antibody (ADA) | Up to 104 weeks
Number of Participants With Neutralizing Antibody (NAb) | Up to 104 weeks
Serum Concentrations of Mezagitamab During and After Intervention | Pre-dose and at multiple time points post-dose, up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (104):
- United States (23):
  - DCR Montgomery, Montgomery, Alabama
  - Academic Medical Research Institute, Los Angeles, California
  - University of California Irvine, Orange, California
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Bioresearch Partners, Miami, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Bioresearch Partners, Pembroke Pines, Florida
  - DCR Columbus, Columbus, Georgia
  - CARE Institute - Boise Kidney, Boise, Idaho
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - DCR Edina, Edina, Minnesota
  - Clinical Research Consultants a JCCT Company, Kansas City, Missouri
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Dallas Renal Group, Dallas, Texas
  - DCR - El Paso, El Paso, Texas
  - Houston Methodist Research Institute - Department of Medicine, Houston, Texas
  - Provecta Research Network, Houston, Texas
  - Nephrology Associates of Houston PLLC, Katy, Texas
  - Sun Research Institute, San Antonio, Texas
  - DCR San Antonio, San Antonio, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia
- Argentina (2):
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (2):
  - Core Research Group, Milton, Queensland
  - Western Health Sunshine Hospital, St Albans, Victoria
- Johannes Kepler Universitat Linz, Universitatsklinik fur Innere 2, Linz, Austria
- China (18):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Changping, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Third Xiangya Hospital of Central South University Yuelu District, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Shandong University - Qilu Hospital, Jinan, Shandong
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Renji Hospital - Eastern Branch, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - The Second Affiliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
- France (3):
  - Hospital Henri Mondor, Créteil, Paris
  - Centre Hospitalier Universitaire de Montpellier (CHU Montpellier) - Hopital Lapeyronie, Montpellier
  - CHU de Nantes, Nantes
- Universitaetsklinikum Jena, Jena, Thuringia, Germany
- The University of Hong Kong - Department of Medicine, Hong Kong, Hong Kong Island, Hong Kong
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Maugeri IRCCS Pavia, Pavia
- Japan (20):
  - Kasugai Municipal Hospital, Kasugai-Shi, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - National Hospital Organization Chiba Medical Center Chibahigashi National Hospital, Chiba, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Toranomon Hospital Kajigaya, Kawasaki-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Japan Community Health care Organization Sendai Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Nara Prefecture General Medical Center, Nara, Nara
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Medical Research Institute KITANO HOSPITAL, PIIF Tazuke-Kofuka, Osaka, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi
- Malaysia (4):
  - Universiti Kebangsaan Malaysia (UKM) - Medical Centre (Pusat Perubatan) (Hospital Canselor Tuanku Muhriz (HCTM)), Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Sultan Idris Shah Serdang (Hospital Serdang), Kajang, Selangor
  - Sunway Medical Centre (SMC), Subang Jaya, Selangor
- Sint Antonius ziekenhuis Utrecht/Nieuwegein, Nieuwegein, Netherlands
- Norway (5):
  - Akershus University Hospital, Lorenskog, Akershus
  - Haukeland Universitetssjukehus, Bergen
  - Sykehuset Ostfold, Grålum
  - Stavanger Universitetssjukehus - Helse Stavanger HF, Stavanger
  - Universitetssykehuset I Trondheim - St. Olavs Hospital - Nevroklinikken, Trondheim
- Poland (2):
  - Nowy Szpital Sp Zo.o, Gmina Świecie
  - SCM Sp. z o.o, Krakow
- Singapore (3):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - National University Hospital, Singapore
- South Korea (3):
  - Ajou University Hospital-Primary Research Location, Suwon, Gyeonggido
  - Seoul National University Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
- Hospital Universitario Virgen del Rocio - PPDS, Seville, Spain
- University Hospital Zurich, Zurich, Switzerland
- Taiwan (5):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Zhongzheng
- United Kingdom (6):
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London, Greater London
  - Birmingham Heartlands Hospital, Birmingham
  - Kent & Canterbury Hospital, Canterbury, Canterbury
  - Hull University Teaching Hospitals NHS Trust, Hull
  - St George's University Hospitals NHS Foundation Trust, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/b04932704fbe42a8??page=1&idFilter=TAK-079-3001